CLINICAL TRIAL: NCT03383341
Title: What's Hopping? Edible Cricket (Gryllodes Sigillatus) Consumption and Gut Microbiota in Healthy Adults, a Double-blind, Randomized Crossover Trial
Brief Title: What's Hopping? Cricket Protein and Human Gut Microbiota
Acronym: HOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Colorado State University (Other)
Collaborators: University of Wisconsin, Madison (Other)
Responsible Party: Principal Investigator, Tiffany Weir, Associate Professor, Colorado State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: 16-6966H
Record Dates: First submitted 2017-12-14; First posted 2017-12-26 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: gut microbiota; cricket powder; prebiotic fiber; inflammation; dietary intervention
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: Randomized, placebo controlled crossover dietary intervention
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Recipes containing cricket powder were matched for taste, color, and texture to creat placebo intervention foods. All foods were prepared by study personnel and then blinded by a third party individual that was not directly associated with the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cricket powder protein (Experimental): Participants were provided with frozen 70 gram breakfast muffins and pre-mixed powder packets to prepare smoothies. Participants were asked to consume one muffin package and one smoothie (mixed with water or choice of milk/milk substitutes) daily for 14 days. The amount of intervention food consumed daily contained 25 grams of cricket protein powder.
  Interventions: Dietary Supplement: Cricket Protein Powder
- Placebo Control (Placebo Comparator): Participants were provided with a placebo comparator that included frozen 70 gram breakfast muffins and pre-mixed powder packets to prepare smoothies. Participants were asked to consume one muffin package and one smoothie (mixed with water or choice of milk/milk substitutes) daily for 14 days. These foods were formulated to taste and appear similar to the cricket intervention foods but did not consume any cricket powder.
  Interventions: Other: Placebo control

INTERVENTIONS:
Dietary Supplement: Cricket Protein Powder — Cricket powder was supplied by Entomo farms and consists of roasted and milled whole crickets.
  Arms: Cricket powder protein
Other: Placebo control — Placebo controls consisted of intervention foods (muffin and smoothie powder packet) that were visually and organoleptically similar to cricket-containing foods but contained no cricket powder.
  Arms: Placebo Control

SUMMARY:
Edible insects are often considered a nutritious, protein-rich, environmentally sustainable alternative to traditional meat. They represent a new food for North American consumers. While the nutrient composition of several insects is characterized, all potential health impacts have not been evaluated. Crickets contain chitin and other fibers that may influence gut health. In this study, we evaluated the effects of consuming 25 grams/day whole cricket powder on gut microbiota composition, while assessing safety and tolerability. Twenty healthy adults participated in this six-week, double-blind, crossover dietary intervention. Participants were randomized into two treatment arms and consumed either cricket-containing or control breakfast foods for 14 days, followed by a 14-day washout period and assignment to the opposite arm. Blood and stool samples were collected at baseline and after each treatment period to assess liver function and microbiota changes. Results demonstrate that cricket consumption is tolerable and non-toxic at the treatment dose. Cricket powder supported growth of the probiotic bacteria, Bifidobacterium animalis, which increased more than 5.7-fold. Cricket consumption was also associated with reduced plasma TNF-a. These data suggest that eating crickets may improve gut health and reduce systemic inflammation; however, more research is needed to understand these effects and underlying mechanisms.

DETAILED DESCRIPTION:
Although no research on the impact of edible insect protein powder on the human microbiome, there is plenty of evidence that edible insects offer a good source nutrition. Extensive research demonstrates that edible insects provide a source of high-quality bioavailable animal protein as many edible insects contain all essential amino acids for human nutrition and have high crude protein levels containing between 40 and 75% protein by dry weight. House crickets, for example, have more protein by dry weight than ground beef or broiled cod fish. Insects are also rich in healthy fatty acids, B vitamins (riboflavin, pantothenic acid, biotin, and folate, as well as important minerals such as iron and zinc. In addition to their nutrient content, and as arthropods, edible insects are also rich in dietary fiber, including chitin, which is found in the exoskeleton.

Chitin is a modified polysaccharide containing nitrogen; it is considered an insoluble fiber with potential prebiotic properties that could benefit human health by selectively promoting the growth of beneficial bacterial species in the intestines. Previous studies on the impact of chitin-glucan derived from Aspergillus niger mycelium on oxidized low-density lipoprotein (OxLDL) in adults, a risk factor for atherosclerosis, found that chitin-glucan intakes of 4.5g/day significantly reduced OxLDL in 6 weeks. Additionally, a study of chito-oligosaccharides found that chitosan derivatives from shrimp cells with a great content of acetylated residues did not cause a putatively prebiotic effect in human gut microbiota-although this study was conducted on human fecal microbiota in batch cultures (not in humans). To date, no comprehensive study has evaluated the impact of whole insect consumption on the microbiota in humans, which would include consumption of insect-derived dietary fibers and chitins with potential health benefits. An assessment of the tolerability of whole insect consumption is also needed, despite the fact that around 2 billion people consume insects on a regular basis in 130 countries or more.

The "What's Hopping? Cricket Protein and Human Gut Microbiota" study will determine the impact of a commercially available insect flour, containing high levels of protein and dietary fiber on human gut bacterial composition and functional capacity. A secondary aim is to establish whether insect powder acts as a prebiotic. In this study, a 100% insect-based flour/powder derived from edible crickets (Acheta domesticus) will be assessed. The objective of this study is to determine if Insect powder consumption changes gut bacteria and reduces inflammation in your intestinal tract compared to a placebo. To this end, we intend to enroll 20 healthy individuals to participate in a crossover diet intervention study. Participants will consume meals made with cricket powder and placebo meals daily for 2 weeks per treatment arm with a 2-week washout period. Both study participants and study personnel (clinical coordinators, PI's, statisticians) will be blinded to the intervention group. Anthropometric measures, as well as stool and blood samples, will be collected at each of 3 clinic visits (baseline, and the end of each intervention period). Primary outcome measures will include gut microbiota and microbial metabolism (determined by measuring fecal short chain fatty acids), local and systemic inflammatory markers, comprehensive metabolic panels and GI health questionnaires to assess safety and tolerability of the intervention foods.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy males and non-pregnant or lactating healthy females of any race or ethnicity and between the ages of 18-65 with a BMI between 18.5-29.9.

Exclusion Criteria:

* Individuals younger than 18 years of age or older than 65 years, and those outside of the BMI range of 18.5-29.9 will be excluded. Individuals will also be excluded if they have taken antibiotics or commercial probiotic/prebiotic supplements within two months of the start of the study treatment. Subjects who self-report food allergies will be excluded from the study because some proteins in insect foods are similar to those found in shellfish that could trigger an allergic reaction and tree nut or dairy products may be used in the breakfast foods.

Additionally, current medications and dietary supplements will be assessed on a case by case basis and will result in exclusion if there is a possibility that the drugs or supplements used would influence the endpoints of the study. This would include statins, metformin, non-steroidal anti-inflammatory drugs (NSAID), Monoamine oxidase inhibitors (MAOI), and botanical supplements that target the gastrointestinal tract or gut microbiota. Individuals with current diagnosis of cancer, liver or kidney disease, gastrointestinal diseases, and metabolic disorders will also be excluded. Pregnant and breastfeeding women will be excluded from the study as well. Additionally, exclusion will be determined if the individual feels they are unable to adhere to the study requirements which include consuming 1 prepared breakfast per day (treatment or placebo) for a total of 28 days (treatment periods), making 3 clinic visits, and providing 3 blood and stool samples.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-05-10 (Actual); Study Completion 2017-05-10 (Actual)

PRIMARY OUTCOMES:
Change in gut microbiota with intervention foods | T=0; Baseline visit prior to starting diet intervention, T1: End of Treatment 1 (2-weeks after the start of intervention), T2: End of study (approximately 6-weeks after T=0 and 2-weeks after starting treatment 2.
  Characterization of microbes in fecal samples using 16s sequencing methodologies.

SECONDARY OUTCOMES:
Change in liver function with intervention foods | T=0; Baseline visit prior to starting diet intervention, T1: End of Treatment 1 (2-weeks after the start of intervention), T2: End of study (approximately 6-weeks after T=0 and 2-weeks after starting treatment 2.
  Comprehensive metabolic panel
Tolerability of intervention foods based on change in GI symptoms | T=0; Baseline visit prior to starting diet intervention, T1: End of Treatment 1 (2-weeks after the start of intervention), T2: End of study (approximately 6-weeks after T=0 and 2-weeks after starting treatment 2.
  Self assessment of gastrointestinal symptoms determined by completion of a questionnaire
Change in mucosal immunity with intervention foods | T=0; Baseline visit prior to starting diet intervention, T1: End of Treatment 1 (2-weeks after the start of intervention), T2: End of study (approximately 6-weeks after T=0 and 2-weeks after starting treatment 2.
  ELISA analysis of secretory Immunoglobulin A (sIgA) in stool samples
Change in microbial metabolism with intervention foods | T=0; Baseline visit prior to starting diet intervention, T1: End of Treatment 1 (2-weeks after the start of intervention), T2: End of study (approximately 6-weeks after T=0 and 2-weeks after starting treatment 2.
  Gas Chromatography determination of fecal short chain fatty acids
Change in lipid metabolism with intervention foods | T=0; Baseline visit prior to starting diet intervention, T1: End of Treatment 1 (2-weeks after the start of intervention), T2: End of study (approximately 6-weeks after T=0 and 2-weeks after starting treatment 2.
  Liquid Chromatography determination of fecal secondary and primary bile acids
Change in systemic inflammation with intervention foods | T=0; Baseline visit prior to starting diet intervention, T1: End of Treatment 1 (2-weeks after the start of intervention), T2: End of study (approximately 6-weeks after T=0 and 2-weeks after starting treatment 2.
  Luminex panel to examine 13 circulating cytokines (pro and anti-inflammatory)

OTHER OUTCOMES:
Change in lipid absorption with intervention foods | T=0; Baseline visit prior to starting diet intervention, T1: End of Treatment 1 (2-weeks after the start of intervention), T2: End of study (approximately 6-weeks after T=0 and 2-weeks after starting treatment 2.
  Colorimetric measure of fecal triglycerides

CONTACTS AND LOCATIONS:
Locations (1):
- Colorado State University, Fort Collins, Colorado, United States

REFERENCES:
- [Result] Stull VJ, Finer E, Bergmans RS, Febvre HP, Longhurst C, Manter DK, Patz JA, Weir TL. Impact of Edible Cricket Consumption on Gut Microbiota in Healthy Adults, a Double-blind, Randomized Crossover Trial. Sci Rep. 2018 Jul 17;8(1):10762. doi: 10.1038/s41598-018-29032-2. PMID 30018370